CLINICAL TRIAL: NCT03943485
Title: Does Implementation of a Uterine Manipulator Prevent Vaginal Length and Sexual Funcation After Abdominal Hysterectomy
Brief Title: Utilization of Uterine Manipulator in Abdominal Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Huseyin Kiyak, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Huseyin1
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Sexual Function Disturbances
Keywords: abdominal hysterectomy; uterine manipulator; vaginal length; sexual function; surgeons' satisfaction
MeSH Terms: conditions — Sexual Dysfunctions, Psychological

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uterien Manipulator Arm (Active Comparator): Patients in this group will receive a uterine manipulator during abdominal hysterectomy.
  Interventions: Device: The uterine manipulator which is primarily used in laparoscopic hysterectomy to accurately locate the colpotomy site. We adopted this device in abdominal hysterectomy.
- Control (No Intervention): Patients in this group will receive standard abdominal hysterectomy without adoption of a uterine manipulator.

INTERVENTIONS:
Device: The uterine manipulator which is primarily used in laparoscopic hysterectomy to accurately locate the colpotomy site. We adopted this device in abdominal hysterectomy. — The uterine manipulator is primarily used in laparoscopic hysterectomy to accurately locate the colpotomy site. We hypothesized that adoption of a uterine manipulator would help the surgeon to better identify the colpotomy site by moving the uterus cranially and thus providing better visualization of the colpotomy site.
  Arms: Uterien Manipulator Arm

SUMMARY:
The investigators aimed to investigate whether the uterine manipulator which is usually utilized in laparoscopic hysterectomy would also be of benefit in preventing postoperative vaginal length and sexual function by facilitating the accurate localization fo the colpotomy site. Patients scheduled for abdominal hysterectomy for benign causes will be randomized into two arms: Group 1 Uterine manipulator arm in which participants received a uterine manipulator during the procedure for aiding to locate the accurate colpotomy site and Group 2 consisting of control patients who will not receive uterine manipulator but undergo a standard abdominal hysterectomy. Postoperative vaginal length, postoperative female sexual function index (FSFI) will be compared with the preoperative measurements in the two groups. A 5 points Surgeon satisfaction scale will also be applied to the surgeons and residents performing the surgery to address their satisfaction in locating the colpotomy site.

DETAILED DESCRIPTION:
The uterine manipulator is a device that facilitates to locate the colpotomy site and visualization of surgical are during laparoscopic hysterectomy. The investigators consider that adoption of the uterine manipulator will also facilitate to locate the colpotomy site in abdominal hysterectomy. Therefore the investigators are planning to enroll patients undergoing an abdominal hysterectomy in this study. Patients will be allocated into one of the study groups: Group 1 Uterine manipulator arm in which participants received a uterine manipulator during the procedure for aiding to locate the accurate colpotomy site and Group 2 consisting of control patients who will not receive uterine manipulator but undergo a standard abdominal hysterectomy. All abdominal hysterectomies will be carried out by the same surgeon under general anesthesia. One week before the surgery vaginal length will be measured and the female sexual function index (FSFI) will be obtained from all patients. Following the surgery vaginal length will again be measured at 3 months and the female sexual function index (FSFI) will be obtained from participants by a research staff who is also a gynecologist. Prevalence of postoperative dyspareunia will be asked to the patients at postoperative 3 months. Just after the surgery, a 5 points surgeons' satisfaction scale will also be completed by the surgeons and residents performing the surgery to address their satisfaction in locating the colpotomy site either with the uterine manipulator as in group 1 or by manually guiding as in group 2.

ELIGIBILITY:
Inclusion Criteria:

- Must be scheduled for total abdominal hysterectomy for benign causes Must be premenopausal Must be sexually active

Exclusion Criteria:

- Apical prolapsus Endometriosis Psychiatric disease

Ages: 40 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Vaginal length | Pre- to the postoperative 3 months
  The change in vaginal length
Female sexual function index (FSFI) | Pre- to the postoperative 3 months
  The change in Female sexual function index score. The Female Sexual Function Index (FSFI) is a brief multidimensional scale for assessing sexual function in women. !9 questions concerning the sexual function are asked. The minimum total score is 4 points. A maximum total score of 36 indicates excellent sexual function. Lower score indicate detoriorated sexual function.

SECONDARY OUTCOMES:
Surgeons' satisfaction: Surgeons' satisfation score | Just after the surgery
  Surgeons' satisfation score. Surgeon satisfaction (SS) and resident satisfaction (RS) for determining the adequate colpotomy site will be evaluated at the end of the procedure surgeon's satisfaction score (SSS) which was scored by the surgical team performing the surgery on a five-point Likert scale as follows: 1 = Very difficult/very poor and 5 = Easy/Good (10). The difference in SS and RS between the two groups will also be a secondary outcome of the present study.

CONTACTS AND LOCATIONS:
Overall Officials: Huseyin Kiyak, MD, Principal Investigator — Kanuni Sultan Suleyman Hospital
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Please Enter the State Or Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No